CLINICAL TRIAL: NCT00545324
Title: A 12 Week Multicenter, Open-Label, Randomized, Observational Study Comparing Singulair® 10 Mg As Controller Monotherapy In Adults With Mild Asthma "To Low Dose" Inhaled Corticosteroid Treatment
Brief Title: First Step With Singulair® Therapy (0476-323)
Acronym: FIRST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0476-323; 2007_025
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast; Duration of Therapy

INTERVENTIONS:
Drug: MK0476 (singulair), montelukast sodium / Duration of Treatment: 6 Weeks
Drug: Comparator: Fluticasone / Duration of Treatment: 6 Weeks

SUMMARY:
In adult patients with mild persistent asthma, singulair® 10 mg will be at least as effective as low dose Inhaled Corticosteroids (ICS) in improving asthma symptom control or satisfaction over a 6 week comparison period.

ELIGIBILITY:
Inclusion Criteria:

* First time diagnosis of mild asthma symptoms which requires an antiinflammatory controller medication
* Patients not controlled with short acting beta2 agonist (sab) therapy (requiring more than one treatment per week but less than 7 per week)
* Patients dissatisfied with low dose ics therapy, or patients reluctant to take ics therapy, or patients insufficiently controlled due to non-compliance with low dose ics therapy through out the preceding 6 weeks
* Patient's forced expiratory volume in one second (fev1) is < 80% of predicted value

Exclusion Criteria:

* Patient on combination therapy
* Patient on long acting beta2 agonists
* Patient on using moderate to high doses of ICS. (ICS >250 &micro g/day flovent&reg; or equivalent per day)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2002-09; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Canadian asthma guidelines criteria

SECONDARY OUTCOMES:
Asthma control questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC